CLINICAL TRIAL: NCT07143071
Title: Endovascular Treatment for Acute High-risk Type B Aortic Dissection in Acute VS Subacute Phase: a Prospective, Multicenter, Non-inferior, Parallel Controlled Trial
Brief Title: EndoVascular Aortic Dissection Early vs Delayed
Acronym: EVADE
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Zhihui Dong, Professor, Shanghai Zhongshan Hospital
Other Study IDs: B2024-370(2)R; 2023ZD0504300 (Other Grant/Funding Number: Noncommunicable Chronic Disease-National Science and Technology Major Project)
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Aortic Dissection Type B
Keywords: aortic dissection; endovascular therapy; timing of intervention
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute high-risk type B aortic dissection: Acute (2-14 days) high-risk type B aortic dissection (defined by one or more of the following: aortic maximum diameter >40 mm, primary tear on the lesser curvature, false lumen diameter >22 mm, entry tear >10 mm, aortic diameter growth >5 mm during hospitalization, imaging evidence of visceral malperfusion, haemorrhagic pleural effusion, need for readmission, or recurrent chest pain).
  Interventions: Procedure: Acute Phase; Procedure: Subacute Phase

INTERVENTIONS:
Procedure: Acute Phase — Patients with acute high-risk type B aortic dissection received endovascular treatment in acute phase (2-14days)
Procedure: Subacute Phase — Patients with acute high-risk type B aortic dissection received endovascular treatment in subacute phase (≥14days)

SUMMARY:
This is a prospective, multicenter, non-inferior, parallel-controlled observational study. This study aims to compare clinical outcomes of endovascular treatment for acute high-risk type B aortic dissection in the acute phase versus the subacute phase. No interventions will be imposed on the patients' standard treatment. Patients with acute high-risk type B aortic dissection will be grouped based on the actual timing of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute (2-14 days) high-risk type B aortic dissection.
* Completion of thoracoabdominal aortic CTA before enrollment.
* Ability to understand the study objectives and voluntarily participate, with signed informed consent from the patient or their legal representative.
* Willingness and ability to comply with follow-up visits and study protocols.

Exclusion Criteria:

* Acute complicated type B aortic dissection.
* Traumatic dissection or penetrating aortic ulcer.
* Connective tissue diseases (e.g., Marfan syndrome, Loeys-Dietz syndrome, Ehlers-Danlos syndrome).
* Pregnancy, women of childbearing potential, or breastfeeding.
* Uncontrolled active infection or active vasculitis.
* Unsuitable access vessels or infection at the access site.
* Endovascular repair requiring ≥2 branch reconstructions.
* Prior aortic surgery (open or endovascular).
* Life expectancy <2 years.
* Myocardial infarction or cerebrovascular accident within 4 weeks before enrollment.
* Severe gastrointestinal bleeding, major surgery, myocardial infarction, or uncorrected coagulation dysfunction within 6 weeks before enrollment.
* Other conditions deemed by the investigator to compromise the patient's medical interests or unlikely adherence to the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute (2-14 days) high-risk type B aortic dissection (defined by one or more of the following: aortic maximum diameter >40 mm, primary tear on the lesser curvature, false lumen diameter >22 mm, entry tear >10 mm, aortic diameter growth >5 mm during hospitalization, imaging evidence of visceral malperfusion, haemorrhagic pleural effusion, need for readmission, or recurrent chest pain).
Sampling Method: Probability Sample
Enrollment: 4068 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality rate | 30 days following the operation
  paraplegia, stroke, new entry tear, renal/liver dysfunction, type I/II/R endoleak
30-day complication rate | 30 days following the operation
  access site complications

SECONDARY OUTCOMES:
Adverse events | 12 months following the operation
  rupture, stent-induced new entry, ischemia (renal/limb/intestinal/spinal), endoleak, dissection aneurysm, stroke, venous thrombosis, all-cause death.
aortic remodeling | 12 months following the operation
  aortic diameter growth > 5 mm in 12 months; dissection aneurysm
5-year all-cause mortality rate | 5 years following the operation
  long-term outcome
5-year complication rate | 5 years following the operation
  long-term outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://zsaorta.com